CLINICAL TRIAL: NCT04672564
Title: A Phase 3, Randomized, Multicenter, Placebo-controlled, Double-blind Clinical Study of the Safety and Efficacy of Carrimycin for Treatment of Severe COVID-19 in Hospitalized Patients
Brief Title: Study to Evaluate Safety and Efficacy of Carrimycin for Treatment of Severe Coronavirus Disease 2019 (COVID-19) in Hospitalized Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: sponsor strategy change
Sponsor: Shenyang Tonglian Group CO., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLKLXG202001
Record Dates: First submitted 2020-12-16; First posted 2020-12-17 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Coronavirus Disease 2019
Keywords: Severe Acute Respiratory Syndrome Coronavirus 2; Safety; Novel coronavirus; Carrimycin; Remdesivir
MeSH Terms: conditions — COVID-19 | interventions — carrimycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carrimycin (Experimental): Patients will receive oral dose of 400 mg carrimycin once-daily and SOC for 14 days.
  Interventions: Drug: Carrimycin
- Placebo (Placebo Comparator): Patients will receive oral dose of Placebo once-daily and SOC for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carrimycin — Carrimycin (400 mg) will be given once-daily for 14 days (2 x 200 mg tablets) after a meal, if a patient experiences an eating problem, carrimycin will be taken without food.
  Arms: Carrimycin
Drug: Placebo — Placebo will be given once-daily for 14 days (2 tablets) after a meal, if a patient experiences an eating problem, placebo will be taken without food.
  Arms: Placebo

SUMMARY:
This is a randomized, multicenter, placebo-controlled, double-blind clinical study in patients hospitalized due to severe Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection.

DETAILED DESCRIPTION:
Eligible 300 hospitalized patients with confirmed severe SARS-CoV-2 infection will be randomly assigned (1:1) to receive 14 days treatment of 400 mg carrimycin and standard of care (SOC) or placebo and SOC.

ELIGIBILITY:
Inclusion Criteria:

* Patient with SARS-CoV-2 infection as determined by real time polymerase chain reaction (RT- PCR) or other commercial or public health assay in any specimen taken ≤ 4 days prior to randomization. Onset of symptoms of COVID-19 must be 14 or fewer days prior to randomization. Patient with a second SARS-CoV-2 episode after resolution of the initial infection may be enrolled if the initial infection had clearly resolved, re-infection is reconfirmed by RT-PCR and all other eligibility criteria are met
* Hospitalized patient who requires oxygen supplementation via either low-flow oxygen device (such as nasal cannula or face mask), high flow oxygen therapy (including high-flow nasal cannula), or non invasive ventilation to maintain peripheral oxygen saturation of at least 94%. The patient must have had such an oxygen requirement for 2 days or fewer at the time of Screening, and the oxygen requirement must be non-improving (worsening or stable) in the Investigator's judgement at the time of Screening and randomization
* Female patient of childbearing potential and male patient with female partner of childbearing potential must agree to use at least one primary form of contraception for the duration of the study
* Ability to provide informed consent personally, or by a legally acceptable representative if the patient is unable to do so
* Patient is willing and able to comply with all required study visits and follow up required by the protocol
* Patient must agree not to enroll in another study of an investigational agent prior to completion of Day 60 of study

Exclusion Criteria:

* Non-hospitalized patients, including those requiring home oxygen support
* Patient has a creatinine clearance < 50 mL/min/1.73m^2 using the modification of diet in renal disease formula
* Patient cannot take the study drug by mouth and needs to be administered by nasogastric tube at Screening.
* Patient has a known allergy to any study medication or macrolides
* Patient with known medical history of hepatitis B or, if tested, presence of hepatitis B surface antigen at Screening
* Patient has a known medical history of hepatitis C or positive hepatitis C antibody test result at Screening (if obtained)
* Patient has a positive hepatitis C RNA test result at Screening
* Patient has a known medical history of human immunodeficiency virus (HIV) infection or was seropositive for human immunodeficiency virus (if tested)
* Patient has been treated with anti-tumor therapy with immunosuppressive effects, which includes chemotherapy, biologics and hormonal therapy in the past 30 days prior to Screening
* Patient has used a macrolide in the week prior to Screening
* Patient has used antiviral drugs which are not part of SOC < 24 hours prior to Day 1
* Patient receiving hemoperfusion or with anticipated use of hemoperfusion (including when hemoperfusion is a part of SOC)
* Patient has used the following types of medications < 2 days prior to Day 1 and/or plans to initiate such medications during the treatment period without an appropriate alternative therapy:

  1. Narrow therapeutic index substrates of cytochrome P450 (CYP) enzymes
  2. Narrow therapeutic index substrates of major transporters: organic anion transporting polypeptide 1B1 and 1B3 (OATP1B1, OATP1B3), organic anion transporter 1 and 3 (OAT1, OAT3), organic cation transporter 2 (OCT2) and multidrug and toxin extrusion proteins 1 and 2-K (MATE1, MATE2K)
  3. Strong inhibitors and/or inducers of enzymes CYP1A2, CYP2B6, CYP2C8, CYP2C9, CYP2C19, CYP2D6, CYP3A4/5
  4. Strong inhibitors of transporters OATP1B1 and OATP1B3
  5. Note: strong inhibitors of OAT1/OAT3, OCT2 and MATE1/MATE2K should be avoided when possible, but when unavoidable investigators may assess the risks and benefits and to continue treatment with such medications under close observation for adverse events
* Patient has consumed foods and/or used herbal medicines with strong CYP3A4 or CYP3A5 effects
* Patient who, in the judgment of the Investigator, will be unlikely or unable to comply with the requirements of this protocol through Day 60
* Female patient who is pregnant or breastfeeding
* Critical patient with a life expectancy < 48 hours
* Patient who has received an organ transplant in the past 6 months prior to Screening or is on the waiting list for organ transplantation
* Patient with evidence of multiorgan failure (defined as two or more organs failing) or septic shock
* Patient requiring mechanical ventilation or extracorporeal membrane oxygenation at Screening
* Patient has a mean corrected QT interval using Fridericia's formula (QTcF) of > 450 msec (for male patients) and > 470 msec (for female patients) at Screening
* Patient who has a history of alcohol abuse within 3 months prior to the study as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Time to patient not requiring supplemental oxygen up to 28 days after randomisation | Up to Day 28
  To evaluate the efficacy of carrimycin with SOC compared to placebo with SOC in patients hospitalized with severe SARS-CoV-2 pneumonia. Patients must have remained off of supplemental oxygen for at least 48 hours and remain off of oxygen until Day 28

SECONDARY OUTCOMES:
Time to recovery based on 8-category ordinal scale | From screening Day (Day -4 to Day -1) until Day 28
  To describe the difference in time to pre-defined symptom improvement compared to placebo, based on 8-category ordinal scale. Time to recovery is defined as time point when a patient reaches level 3 or lower on the 8-Category ordinal scale and does not return to a level > 3 during the 28-day period. The 8-Category ordinal scale score ranges from 1 to 8. Score 1: Not hospitalized, no limitations on activities; 2: Not hospitalized, limitation on activities, home oxygen requirement or both; 3: Hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care; 4: Hospitalized, not requiring supplemental oxygen but requiring ongoing medical care; 5: Hospitalized, requiring supplemental oxygen; 6: Hospitalized, requiring noninvasive ventilation or high flow oxygen devices; 7: Hospitalized, receiving invasive mechanical ventilation or extracorporeal membrane oxygenation and score 8: Death. Higher scores indicate worse outcome.
Time to recovery based on the Breathlessness, Cough and Sputum Scale (BCSS) | From screening Day (Day -4 to Day -1) until Day 28
  To describe the difference in time to pre-defined symptom improvement compared to placebo based on the BCSS. The BCSS is a three-item questionnaire rating breathlessness, cough and sputum on a 5-point Likert scale from 0 (no symptoms) to 4 (severe symptoms). A reduction in the mean total BCSS score represents a substantial symptomatic improvement.
Time to symptom improvement | From screening Day (Day -4 to Day -1) until Day 28
  To describe the difference in time to pre-defined symptom improvement compared to placebo, based on the BCSS. Time to symptom improvement can be considered when the score of a patient has a reduction of 1 with 2 consecutive ratings on the BCSS. The BCSS is a three-item questionnaire rating breathlessness, cough and sputum on a 5-point Likert scale from 0 (no symptoms) to 4 (severe symptoms). A reduction in the mean total BCSS score represents a substantial symptomatic improvement.
Length of hospital stay (in days) | From Screening Day (Day -4 to Day -1) until Day 60 or Early Withdrawal
  To evaluate length of hospital stay between patients receiving carrimycin vs placebo.
Time to discharge (in days) | From screening Day (Day -4 to Day -1) until Day 60 and at Early Withdrawal
  To evaluate time to discharge between patients receiving carrimycin vs placebo.
Number of patients with all cause mortality at Days 14 and 28 | At Days 14 and 28
  To evaluate mortality rates between patients receiving carrimycin vs placebo.
Changes from baseline in sequential organ failure assessment (SOFA) score | From baseline (Day -4 to Day -1) Days 3, 7, 10, 14 and 28 after treatment
  To evaluate the improvement for specific clinical parameters including fever, respiratory rate, oxygen saturation, breathlessness, cough and sputum production. The SOFA score ranges from 0 to 4. Lower score predicts better organ functioning and higher score represents severe organ failure.
Percentage of patients who reach level 2 or lower at Day 28 on the 8 category ordinal scale | From screening Day (Day -4 to Day -1) until Day 28
  The 8-Category ordinal scale score ranges from 1 to 8. Score 1: Not hospitalized, no limitations on activities; 2: Not hospitalized, limitation on activities, home oxygen requirement or both; 3: Hospitalized, not requiring supplemental oxygen and no longer requiring ongoing medical care; 4: Hospitalized, not requiring supplemental oxygen but requiring ongoing medical care; 5: Hospitalized, requiring supplemental oxygen; 6: Hospitalized, requiring noninvasive ventilation or high flow oxygen devices; 7: Hospitalized, receiving invasive mechanical ventilation or extracorporeal membrane oxygenation and score 8: Death. Higher scores indicate worse outcome.
Mean changes in BCSS score during the study period | From screening Day (Day -4 to Day -1) until Day 28
  To evaluate the improvement for specific clinical parameters including breathlessness, cough and sputum production. The BCSS is a three-item questionnaire rating breathlessness, cough and sputum on a 5-point Likert scale from 0 (no symptoms) to 4 (severe symptoms). A reduction in the mean total BCSS score represents a substantial symptomatic improvement.
Change from baseline in respiratory rate | From screening Day (Day -4 to Day -1) until Day 60 and at Early Withdrawal
  To evaluate the improvement for specific clinical parameters including respiratory rate.
Change from baseline in temperature | From screening Day (Day -4 to Day -1) until Day 60 and at Early Withdrawal
  To evaluate the improvement for specific clinical parameters including fever.
Number of patients with adverse event (AEs) and Serious adverse events (SAEs) | From screening Day (Day -4 to Day -1) until Day 28 and until Day 60
  To evaluate the safety and tolerability of the carrimycin and to describe the safety profile of treatments as reflected by AEs and SAEs.

CONTACTS AND LOCATIONS:
Locations (17):
- PharmaTex Research, LLC, Amarillo, Texas, United States
- Instituto Médico Platense, La Plata, Buenos Aires, Argentina
- Brazil (2):
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto - Hospital de Base, São José do Rio Preto, São Paulo
- Mexico (3):
  - Nuevo Hospital Civil de Guadalajara "Juan I. Menchaca", Guadalajara, Jalisco
  - EME RED Hospitalaria, Mérida, Yucatán
  - Hospital Dr. Agustin O'Horan, Mérida, Yucatán
- Philippines (5):
  - St. Paul's Hospital of Iloilo, Inc., Iloilo City, Iloilo
  - Makati Medical Center - Infectious Diseases, Makati City, National Capital Region
  - San Juan De Dios Hospital, Pasay, National Capital Region
  - Veterans Memorial Medical Center, Quezon City, National Capital Region
  - Quirino Memorial Medical Center, Quezon City, National Capital Region
- Ukraine (5):
  - Chernihivska miska likarnia #2, Chernihiv, Chernihiv Oblast
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Oblasnyi klinichnyi ftyziopulmonolohichnyi tsentr, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Komunalne Pidpryiemstvo "Poltavska Oblasna Klinichna Infektsiina Likarnia" Poltavskoi Oblasnoi Rady, Poltava, Poltava Oblast
  - Volyn Regional Clinical Hospital, Lutsk, Volyn Oblast